CLINICAL TRIAL: NCT06351787
Title: Cortical Activity of a Body Scan Meditation and Yoga Practice in Healthy Adults: Correlates With Interoceptive Awareness, Healthy Emotionality, and Pain Perception
Brief Title: Project Soma: Cortical Activity of a Body Scan Meditation and Yoga Practice in Healthy Yogis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 22-X-97
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Well-Being, Psychological
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: A 2-armed randomized cross-sectional experimental study with 20 healthy participants who hold yoga experience.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Body scan (Experimental): Participants will follow an audio-guided meditation in the sitting posture, which provides systematic verbal cues to draw their attention to different body parts to cultivate non-judgmental awareness. This will be performed in blocks of 2-minute increments, for up to 10 minutes, interspersed with 30-second periods of rest - where the participant will allow their mind to wander freely.
  Interventions: Behavioral: Resting and movement-based focused awareness meditations
- Yoga (Experimental): Participants will follow a video-guided yoga session in the standing posture, which provides verbal and visual cues to draw their attention to their body and breath during upright yoga postures. This practice occurs in 2-minute active intervals for up to 10 minutes, interspersed with 30-second rest to be consistent with the experimental block design.
  Interventions: Behavioral: Resting and movement-based focused awareness meditations

INTERVENTIONS:
Behavioral: Resting and movement-based focused awareness meditations — Resting and movement-based focused awareness meditations

SUMMARY:
In this 2-armed randomized cross-sectional experimental study of healthy participants with yoga experience, we will examine the relationship between 4 self-reported enhancing psychological factors, cortical activity captured with functional near-infrared spectroscopy (fNIRS), and pain sensitivity (mechanical pressure pain tolerance) captured with algometry.

Specifically, we will examine the correlates of interoceptive awareness and mindful awareness with cortical activity (Aim 1a) and pain tolerance (Aim 1b); determine cortical activity responsiveness of two brief awareness-focused meditations - a resting-based body scan practice and yoga practice (Aim 2a); characterize cortical activity profiles with sequentially delivered body scan and yoga practices (Aim 2b); and elucidate the relationship between interoceptive awareness with healthy emotionality and psychological wellbeing (Aim 3).

Our central hypotheses are that (Aim 1a) higher interoceptive awareness and mindful awareness will moderately correlate with higher cortical activity for both awareness-focused meditation practices; (Aim 1b) individuals sub-grouped into the 'acceptance in action cluster' based on 2 self-report measures will exhibit higher pain tolerance; (Aim 2a) cortical activity will be higher in the yoga practice compared to the body scan practice; and (Aim 2b) higher cortical activity will be observed in the body scan->yoga intervention sequence compared to the yoga->body scan intervention sequence. Furthermore, (Aim 3) we predict that interoceptive awareness will moderately correlate with healthy emotionality and psychological well-being.

DETAILED DESCRIPTION:
In Aim 1a, we will use self-report measures of interoception and awareness, using the Multidimensional Assessment of Interoceptive Awareness (MAIA) and the Five Facet Mindfulness Questionnaire - Short Form (FFMQ-SF), and fNIRS to capture cortical activity during brief exposures to resting (Body scan) and movement-based (yoga) practices. We predict that self-reported interoception and awareness will moderately, and directly correlate with prefrontal cortical activity during the Body Scan and Yoga practices. In other words, we expect that higher levels of self-reported interoception and awareness will be positively associated with higher levels of prefrontal cortical activity for both awareness-focused practices.

In Aim 1b, we will use (i) the self-report measures (MAIA and FFMQ-SF) to identify a 'regulatory awareness' cluster and 'acceptance in action' cluster, and (ii) the quantitative sensory test of pressure pain tolerance. We will test the hypothesis that individuals categorized into the 'acceptance in action' cluster will demonstrate higher pressure pain threshold and tolerance compared to the 'regulatory awareness' cluster.

In Aim 2, we will use cortical activity levels captured using fNIRS during two awareness-based practices - Body Scan and Yoga. We expect that cortical activity will be higher during Yoga compared to Body Scan (Aim 2a). We further expect that individuals who initially receive the resting-based meditation and then progress to receive the active-based meditation (Body Scan->Yoga) will at a group level demonstrate higher levels of cortical activity in comparison to individuals who receive Yoga->Body Scan (Aim 2b).

In Aim 3, we will use self-report measures of interoception (MAIA) and self-report measures of healthy emotionality (Emotional Styles Questionnaire, ESQ) and psychological well-being (Scales of Psychological Well-Being, PWB). We predict that interoception will be moderately correlated with healthy emotionality and psychological well-being.

Our contribution will be significant because elucidating cognitive and affective processes of awareness-based practices will help inform who may more favorably respond to different awareness-based practices aimed at cultivating well-being. Our proposed research is innovative because it seeks to advance a sensorimotor and psychological mechanistic understanding of meditation practices that will elucidate the 'active ingredients' responsible for its therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

* Adults currently engaged in yoga

Exclusion Criteria:

* History of any neurological disorder that could impair brain function

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Cortical activity | Baseline (T0)
  Oxy-Hb and De-Oxy-Hb
Interoceptive awareness | Baseline (T0)
  Multidimensional Assessment of Interoceptive Awareness (MAIA)
Mindful awareness | Baseline (T0)
  Five Facet Mindfulness Questionnaire - Short form (FFMQ-SF)
Pressure pain threshold and tolerance | Baseline (T0)
  Computerized pressure pain algometry applied over the ventral thenar eminence, 3 series of ascending stimulus intensities, applied as a slowly increasing ramp of 50 kPa/s. Pain threshold is defined as the first perception or detection of pain, or a numeric rating of 2 on a scale of 0 to 10, where 0 = no sensation and 10 = worst imaginable pain. Pain tolerance is defined as the point of maximum tolerable pain, a numeric pain rating of 8 on a scale of 0 to 10.

SECONDARY OUTCOMES:
Healthy emotionality | Baseline (T0)
  Emotional Styles Questionnaire (ESQ)
Well-being | Baseline (T0)
  Scales of Psychological Well-Being (SPWB)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Karayannis, Principal Investigator — Ohio University
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided